CLINICAL TRIAL: NCT04465981
Title: A Longitudinal, Non-randomized Study to Evaluate the Utility of the INanoBio's Protein Arrays in Detecting Unique Antibodies in COVID-19 Patients
Brief Title: Investigation of Antibody and Immune Responses to SARS-CoV-2 Proteins in COVID-19 Patients
Acronym: SARS-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: INanoBio Inc. (Industry)
Collaborators: TMC HealthCare (Other)
Responsible Party: Sponsor
Other Study IDs: INANO-CV1
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum will be isolated from periodic clinical blood specimens during the entire duration of the patient's hospital stay. Whole blood and plasma may also be collected. The CoV-2 protein serology assay will be performed on each sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with lab-confirmed COVID-19: Subject has lab-confirmed diagnosis of COVID-19 by RT-PCR
  Interventions: Diagnostic Test: Sampling
- Patients who are suspected to have or are confirmed to not have COVID-19: Subject has suspected COVID-19 according to medical evaluation, but does not yet have lab-confirmed diagnosis of COVID-19 (results outstanding, or has tested negative by RT-PCR)
  Interventions: Diagnostic Test: Sampling

INTERVENTIONS:
Diagnostic Test: Sampling — Test is to validate the utility of INanoBio's automated protein arrays in detecting antibodies against SARS-CoV-2 proteins.

SUMMARY:
SARS-CoV-2, the virus that causes coronavirus disease 2019 (COVID-19), has negatively impacted global health and requires more research to develop better tests and to improve disease treatment.

The purpose of this research is to aid in the testing effort by collecting samples from people who have been diagnosed with COVID-19 or are suspected of having COVID-19. Samples you provide will be used investigationally by INanoBio to develop a test to determine when antibodies against various SARS-CoV-2 proteins are detectable.

Up to approximately 80 subjects of all ages with either a suspected or lab-confirmed diagnosis of COVID-19 will take part in this research.

DETAILED DESCRIPTION:
A longitudinal, non-randomized study to evaluate the utility of the INanoBio's protein arrays in detecting unique antibodies in COVID-19 patients. To study the feasibility of utilizing a viral proteome microarray for evaluating exposure status, immunity status, diagnosis, and prognosis of SARS-CoV-2 infections during and after the course of disease. The sample size is to include 80 subjects: 40 diagnosed with COVID-19 and 40 suspected to have COVID-19. The goal will be to assess antibodies throughout the subject's disease course compared to controls.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following criteria to be eligible for treatment in the study:

1. Subject or legal representative understands the nature of the procedure and has signed the Subject Informed Consent Form prior to study procedures
2. For the COVID-19 Cohort

   * Subject has lab-confirmed diagnosis of COVID-19 by RT-PCR
3. For the PUI Cohort

   * Subject has suspected COVID-19 according to medical evaluation, but does not yet have lab-confirmed diagnosis of COVID-19 (results outstanding, or has tested negative by RT-PCR)

Exclusion Criteria:

* Subject or legal representative not willing to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 tested patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Serological identification of individuals who have been infected with SARS-CoV-2 | Through study completion, an average of 1 year
  Distinguish individuals who have been infected with SARS-CoV-2 from those who have not using antibody-based assays and measure antibody levels as a function of time

SECONDARY OUTCOMES:
Identify antibody and/or immune signatures in COVID-19 patients | Through study completion, an average of 1 year
  Analyze and identify antibody and/or immune signatures in COVID-19 patients that differentiate patients with severe disease versus those without, and determine which antigens are most useful for serological testing

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Scott, Principal Investigator — TMC HealthCare
Locations (1):
- TMC HealthCare, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No